CLINICAL TRIAL: NCT03964415
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase 3 Efficacy Study of a Heterologous Vaccine Regimen of Ad26.Mos4.HIV and Adjuvanted Clade C gp140 and Mosaic gp140 to Prevent HIV-1 Infection Among Cis-gender Men and Transgender Individuals Who Have Sex With Cis-gender Men and/or Transgender Individuals
Brief Title: A Study of Heterologous Vaccine Regimen of Adenovirus Serotype 26 Mosaic4 Human Immunodeficiency Virus(Ad26.Mos4.HIV), Adjuvanted Clade C gp140 and Mosaic gp140 to Prevent HIV-1 Infection Among Cis-gender Men and Transgender Individuals Who Have Sex With Cis-gender Men and/or Transgender Individuals
Acronym: MOSAICO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CR108604; 2018-003666-13 (EudraCT Number); VAC89220HPX3002 (Other: Janssen Vaccines & Prevention B.V.); HVTN 706 (Other: HIV Vaccine Trials Network (HVTN))
Record Dates: First submitted 2019-05-24; First posted 2019-05-28 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group1:Ad26.Mos4.HIV,Clade C and Mosaic gp140 bivalent vaccine (Experimental): Participants will receive adenovirus serotype 26.Mosaic 4.human immunodeficiency virus (Ad26.Mos4.HIV) via intramuscular (IM) injection into the deltoid muscle at months 0 (Day 1) and 3 (preferably the deltoid of the non-dominant upper arm) and, Ad26.Mos4.HIV together with Clade C and Mosaic gp140 HIV bivalent vaccine IM into the deltoid muscle at Months 6 and 12 (different deltoid for each injection).
  Interventions: Biological: Ad26.Mos4.HIV; Biological: Clade C and Mosaic gp140 HIV bivalent vaccine
- Group 2: Placebo (Placebo Comparator): Participants will receive placebo into the deltoid muscle on Months 0 (Day 1), 3 (1 injection), 6 and 12 (2 injections).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Ad26.Mos4.HIV — Participants will receive Ad26.Mos4.HIV via IM injection into the deltoid muscle at months 0 (Day 1), 3, 6 and 12.
  Arms: Group1:Ad26.Mos4.HIV,Clade C and Mosaic gp140 bivalent vaccine
Biological: Clade C and Mosaic gp140 HIV bivalent vaccine — Participants will receive Clade C and Mosaic gp140 HIV bivalent vaccine as IM injection into the deltoid muscle at Months 6 and 12.
  Arms: Group1:Ad26.Mos4.HIV,Clade C and Mosaic gp140 bivalent vaccine
Biological: Placebo — Participants will receive matching placebo.
  Arms: Group 2: Placebo

SUMMARY:
The purpose of this study is to evaluate the vaccine efficacy (VE) of a heterologous vaccine regimen utilizing Ad26.Mos4.HIV and aluminum phosphate-adjuvanted Clade C gp140 and Mosaic gp140 for the prevention of HIV-1 infection in HIV-1 seronegative cis-gender men and transgender individuals having sex with cis-gender men and/or transgender individuals.

DETAILED DESCRIPTION:
Human immunodeficiency virus type 1 (HIV-1) is a retrovirus that, if left untreated, can progress to acquired immunodeficiency syndrome (AIDS), a condition in which the immune system is severely compromised, leading to life-threatening conditions. Ad26.Mos4.HIV is a tetravalent vaccine composed of Ad26.Mos1.Gag-Pol, Ad26.Mos2.Gag-Pol, Ad26.Mos1.Env, and Ad26.Mos2S.Env. Clade C and Mosaic gp140 HIV bivalent vaccine contains: Clade C gp140, HIV-1 Env gp140 of Clade C, Mosaic gp140, HIV-1 Env gp140, and aluminum phosphate adjuvant. Evidences showed that a combination of vaccination with Ad26.Mos.HIV followed by Ad26.Mos.HIV together with Clade C gp140 protein in aluminum phosphate adjuvant led to highest level of protection observed so far with this vaccine concept. Study comprises of a screening period of 45 days, a 12-month vaccination period and a follow-up period of at least 18 months after fourth vaccination (until Month 30) in participants who remain HIV-1 negative or up to 6 months after diagnosis of HIV-1 infection in participants who become HIV-1 infected. Participants who completed their Month 30 visit will be followed for HIV infection, medically-attended adverse event (MAAEs) and serious adverse events until the end of study (Month 30). Primary analysis of vaccine efficacy will evaluate the number of HIV-1 infections in the vaccine group compared to number of HIV-1 infections in the placebo group between Month 7 and Month X (with 24<=X<=30) in per-protocol population.

ELIGIBILITY:
Inclusion Criteria:

* Individual is either cis-gender man having sex with cis-gender men and/or transgender individuals or transgender woman having sex with cis-gender men and/or transgender individuals or transgender man having sex with cis-gender men and/or transgender women or gender non-conforming individual having receptive or insertive anal and/or vaginal condom-less intercourse and who is considered by the site staff to be at increased risk for HIV-1 infection. The potential participants must in the last 6 months have had any condom-less receptive anal or vaginal sex (not included is condom-less anal sex within a mutually monogamous relationship >=12 months if the partner is HIV negative or living with HIV and virally suppressed) or rectal or urethral gonorrhea or chlamydia or incident syphilis or any stimulant use or any other drug and/or substance which in the local context may be associated with increased HIV transmission (example, cocaine, amphetamine) or 5 or more sex partners
* Potential participant has a negative test result for HIV-1 and HIV-2 infection less than or equal to (<=) 28 days prior to first vaccination
* Potential participant must be healthy based on medical history, physical examination, and vital sign measurement performed at screening
* Contraceptive use by participants assigned female at birth and who have not had sexual reassignment surgery should be consistent with local regulations regarding the acceptable methods of contraception for those participating in clinical studies
* All participants of childbearing potential must have a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test at screening and have a negative urine beta-hCG pregnancy test immediately prior to each study vaccine administration

Exclusion Criteria:

* Potential participants choosing to use PrEP. However, once participants are enrolled and received their first vaccination, and they change their mind regarding PrEP usage, they will be allowed to take PrEP according to the site PrEP plan and will continue to receive further vaccinations. The use of long acting PrEP is disallowed from 24 months prior to Day 1
* Potential participant is a recipient of a HIV-vaccine candidate at any time, or a recipient of other experimental vaccine(s) within the last 12 months prior to Day 1. For participants who received an experimental vaccine (except HIV vaccine) more than 12 months prior to Day 1, documentation of the identity of the experimental vaccine must be provided to the HPX3002/HVTN 706 safety review team, who will determine eligibility on a case by-case basis. Exceptions: participants can be included if the vaccine received (except HIV vaccine) was subsequently licensed or authorized for emergency use (example, Emergency Use Authorization (EUA), Emergency Use Listing (EUL), or similar program). Participants with proof of having received only placebo can also be included. Participants who are currently still in an interventional study of such a licensed/emergency use-authorized vaccine are to be excluded from the current study
* Potential participant has received an HIV-related mAb, whether licensed or investigational, within the last 12 months prior to Day 1. For participants who received an HIV-related mAb more than 12 months prior to Day 1, documentation of the identity of the mAb must be provided to the HPX3002/HVTN 706 safety review team, who will determine eligibility on a case-by-case basis
* Potential participant has known allergy or history of anaphylaxis or other serious adverse reactions to vaccines
* Pregnant, or breast-feeding, or planning to become pregnant while enrolled in this study or within 90 days after the last dose of study vaccination

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cis-gender men and transgender individuals who have sex with cis-gender men and/or transgender Individuals.
Enrollment: 3900 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (53):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Bridge HIV, San Francisco, California
  - Whitman Walker Health, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Emory University Rollins School of Public Health - Ponce De Leon CRS, Atlanta, Georgia
  - The Hope Clinic at Emory University, Decatur, Georgia
  - University Of Illinois, Chicago, Illinois
  - New Orleans Adolescent Trials Unit CRS, New Orleans, Louisiana
  - Dana-Farber/Brigham and Women's Hospital, Boston, Massachusetts
  - Fenway Health, Boston, Massachusetts
  - Rutgers, The State University of New Jersey - The University Hospital/ACTG Network, Newark, New Jersey
  - Harlem Prevention Center CRS, New York, New York
  - Columbia University Medical Center, New York, New York
  - New York Blood Center, New York, New York
  - Strong Memorial Infectious Disease, Rochester, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Gordon E. Crofoot MD, Houston, Texas
  - Seattle Vaccine Trials Unit, Seattle, Washington
- Argentina (4):
  - Helios Salud Sa, Buenos Aires
  - Fundacion Huesped, Ciudad Autonoma de Buenos Aire
  - Hospital J. M. Ramos Mejía, Ciudad de Buenos Aires
  - Instituto Caici Srl., Rosario
- Brazil (8):
  - Universidade Federal De Minas Gerais - Hospital das Clínicas, Belo Horizonte
  - Centro Medico Sao Francisco, Curitiba
  - Fundacao de Medicina Tropical Doutor Heitor Vieira Dourado - FMT, Manaus
  - Fundacao Oswaldo Cruz, Rio de Janeiro
  - Municipio de Nova Iguacu - Hospital Geral de Nova Iguacu, Rio de Janeiro
  - Instituto de infectologia Emilio Ribas, São Paulo
  - Hospital Das Clinicas Da Faculdade De Medicina Da USP, São Paulo
  - Centro de Referencia E Treinamento Dst/Aids, São Paulo
- Italy (3):
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliero-Universitaria Policlinico di Modena, Modena
  - Istituto nazionale malattie infettive 'L. Spallanzani', Roma
- Mexico (3):
  - Hospital Civil Fray Antonio Alcalde, Guadalajara
  - Inst. Nal. de Ciencias Med. Y Nutricion Salvador Zubiran, Mexico City
  - Unidad de Atención Medica e Investigacion en Salud (UNAMIS), Mérida
- Peru (5):
  - Centro de Investigaciones Tecnologicas, Biomedica y medio ambientales (CITBM), Callao
  - Asociacion Civil Selva Amazonica (ACSA), Iquitos
  - Asociacion Civil Via Libre, Lima
  - Asociacion Civil Impacta Salud y Educacion - Barranco, Lima - Barranco
  - Asociacion Civil Impacta Salud y Educacion- San Miguel CRS, Lima - San Miguel
- Poland (2):
  - Neutrum Lekarze M.Hlebowicz i Partnerzy spolka partnerska, Gdansk
  - Wroclawskie Centrum Zdrowia SPZOZ, Poradnia Profilaktyczno-Lecznicza, Wroclaw
- Puerto Rico (2):
  - Clinical Research Puerto Rico Inc, San Juan
  - University of Puerto Rico, San Juan
- Spain (6):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp. Univ. Vall D Hebron, Barcelona
  - Hosp Reina Sofia, Córdoba
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Hosp. Clinico San Carlos, Madrid
  - Hosp. Gral. Univ. Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Buchbinder SP, Spinosa Guzman S, Sanchez J, Willems W, Stieh DJ, van Duijn J, van Rosmalen MGM, Hendriks J, Nijs S, Lavreys L, Paez CA, Grinzstejn B, Hutter J, Mann P, Sierra Madero JG, Cahn P, Castagna A, Truyers C, Roels S, Gilbert PB, Carone M, Luedtke A, Corey L, Pau MG, Tomaka F; HVTN 706/HPX3002/Mosaico Study Team. Efficacy and safety of a mosaic HIV-1 vaccine regimen in men who have sex with men and transgender individuals (HVTN 706/HPX3002/Mosaico): a global, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet HIV. 2025 Dec;12(12):e823-e835. doi: 10.1016/S2352-3018(25)00195-X. PMID 41314741

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Ad26.Mos4.HIV + Clade C and Mosaic gp140: Participants received adenovirus serotype 26.Mosaic 4.human immunodeficiency virus (Ad26.Mos4.HIV) 5*10^10 viral particles (vp) intramuscular (IM) injection into the deltoid muscle as a monotherapy at Months 0 (Day 1) and 3 (Day 84) (preferably the deltoid of the non-dominant upper arm) along with adjuvanted protein formulation consisting of Clade C protein 80 micrograms (mcg), Mosaic protein 75 mcg and adjuvanted aluminum phosphate 425 mcg, into the deltoid muscle at Months 6 (Day 168) and 12 (Day 364) (different deltoid for each injection).
- Group 2: Placebo: Participants received placebo into the deltoid muscle at Months 0 (Day 1), 3 (Day 84; 1 injection), 6 (Day 168) and 12 (Day 364; 2 injections).
Period: Overall Study
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C and Mosaic gp140 | Group 2: Placebo
Started | 1948 | 1952
Treated: Full Analysis Set (FAS) | 1942 | 1945
Completed | 95 | 103
Not Completed | 1853 | 1849
Not completed — Sponsor's decision | 1563 | 1528
Not completed — Lost to Follow-up | 139 | 146
Not completed — Withdrawal by Subject | 68 | 72
Not completed — Physician Decision | 34 | 48
Not completed — Adverse Event | 3 | 0
Not completed — Death | 4 | 6
Not completed — Protocol Violation | 1 | 4
Not completed — Other | 35 | 38
Not completed — Randomized but not treated | 6 | 7

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) set included all randomized participants who received at least one vaccine administration.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C and Mosaic gp140 | Group 2: Placebo | Total
Number analyzed (Participants) | 1942 | 1945 | 3887
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.7 (8.28) | 29.9 (8.58) | 29.8 (8.43)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female (at birth) | 9 | 7 | 16
  Male (at birth) | 1933 | 1937 | 3870
  Undifferentiated (at birth) | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1690 | 1675 | 3365
  Not Hispanic or Latino | 238 | 246 | 484
  Unknown or Not Reported | 14 | 24 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 63 | 59 | 122
  Asian | 13 | 12 | 25
  Native Hawaiian or Other Pacific Islander | 3 | 7 | 10
  Black or African American | 140 | 161 | 301
  White | 868 | 862 | 1730
  More than one race | 814 | 809 | 1623
  Unknown or Not Reported | 41 | 35 | 76
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 202 | 203 | 405
  Brazil | 425 | 426 | 851
  Italy | 46 | 44 | 90
  Mexico | 175 | 172 | 347
  Peru | 812 | 808 | 1620
  Poland | 57 | 60 | 117
  Puerto Rico | 5 | 5 | 10
  Spain | 128 | 130 | 258
  United States | 92 | 97 | 189

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Confirmed Human Immunodeficiency Virus (HIV)-1 Infections Diagnosed Between the Month 7 and Month 24 Visits (Per-protocol [PP] Set)
Description: Number of participants with a confirmed HIV-1 infections diagnosed between the Month 7 and Month 24 visits (PP set) was reported. The data represents the cumulative incidence of HIV-1 infections.
Time Frame: From Month 7 up to Month 24
Population: The PP set included all participants in the full analysis set (FAS; all randomized participants who received at least one vaccine administration) population who had a negative HIV test 4 weeks post 3rd vaccination visit (that is, at the Month 7 Visit) and who received all planned vaccinations at the first three vaccination visits within the respective visit windows.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C and Mosaic gp140 | Group 2: Placebo
Number analyzed (Participants) | 1525 | 1494
Participants | 65 | 58

2. Primary Outcome: Number of Participants With a Confirmed Human Immunodeficiency Virus (HIV)-1 Infections Diagnosed Between the Month 7 and Month 30 Visits (PP Set)
Description: Number of participants with a confirmed HIV-1 infections diagnosed between the Month 7 and Month 30 visits (PP set) was reported. The data represents the cumulative incidence of HIV-1 infections.
Time Frame: From Month 7 up to Month 30
Population: The PP set included all participants in the FAS (all randomized participants who received at least one vaccine administration) population who had a negative HIV test 4 weeks post 3rd vaccination visit (that is, at the Month 7 Visit) and who received all planned vaccinations at the first three vaccination visits within the respective visit windows.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C and Mosaic gp140 | Group 2: Placebo
Number analyzed (Participants) | 1525 | 1494
Participants | 71 | 67

3. Secondary Outcome: Number of Participants With Solicited Local Adverse Events (AEs)
Description: Number of participants with solicited local AEs were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, are used to assess the reactogenicity of the study vaccine and are pre-defined local (injection site) and which were noted by participants in their participant diary for 7 days post vaccination (day of vaccination and the subsequent 7 days).
Time Frame: Up to 7 days post each vaccination (dose) on Days 1 (up to Day 8), 84 (up to Day 91), 168 (up to Day 175), and 364 (up to 371)
Population: The FAS set included all randomized participants who received at least one vaccine administration. Here, 'n' (number analyzed) is defined as participants analyzed at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C and Mosaic gp140 | Group 2: Placebo
Number analyzed (Participants) | 1942 | 1945
Participants
  Up to 7 days post dose on Day 1 | 1225 | 329
  Up to 7 days post dose on Day 84: number analyzed (Participants) | 1888 | 1877
  Up to 7 days post dose on Day 84 | 905 | 239
  Up to 7 days post dose on Day 168: number analyzed (Participants) | 1841 | 1816
  Up to 7 days post dose on Day 168 | 1010 | 319
  Up to 7 days post dose on Day 364: number analyzed (Participants) | 1724 | 1715
  Up to 7 days post dose on Day 364 | 917 | 252

4. Secondary Outcome: Number of Participants With Solicited Systemic Adverse Events (AEs)
Description: Number of participants with solicited systemic AEs were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited systemic events included events such as fatigue, headache, nausea, and myalgia, for which participants were specifically questioned and which were noted by participants in their participant diary for 7 days post vaccination (day of vaccination and the subsequent 7 days).
Time Frame: Up to 7 days after each vaccination (dose) on Days 1 (up to Day 8), 84 (up to Day 91), 168 (up to Day 175), and 364 (up to 371)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C and Mosaic gp140 | Group 2: Placebo
Number analyzed (Participants) | 1942 | 1945
Participants
  Up to 7 days post dose on Day 1 | 1313 | 860
  Up to 7 days post dose on Day 84: number analyzed (Participants) | 1888 | 1877
  Up to 7 days post dose on Day 84 | 891 | 572
  Up to 7 days post dose on Day 168: number analyzed (Participants) | 1841 | 1816
  Up to 7 days post dose on Day 168 | 856 | 535
  Up to 7 days post dose on Day 371: number analyzed (Participants) | 1724 | 1715
  Up to 7 days post dose on Day 371 | 759 | 432

5. Secondary Outcome: Number of Participants With Unsolicited Adverse Events (AEs)
Description: Number of participants with unsolicited AEs were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs are all AEs for which the participants were not specifically questioned in the participant's diary.
Time Frame: Up to 28 days after each vaccination (dose) on Days 1 (up to Day 29), 84 (up to Day 112), 168 (up to Day 196), and 364 (up to 392)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C and Mosaic gp140 | Group 2: Placebo
Number analyzed (Participants) | 1942 | 1945
Participants
  Up to 28 days post dose on Day 1 | 253 | 245
  Up to 28 days post dose on Day 84: number analyzed (Participants) | 1888 | 1877
  Up to 28 days post dose on Day 84 | 190 | 191
  Up to 28 days post dose on Day 168: number analyzed (Participants) | 1841 | 1816
  Up to 28 days post dose on Day 168 | 298 | 293
  Up to 28 days post dose on Day 364: number analyzed (Participants) | 1724 | 1715
  Up to 28 days post dose on Day 364 | 249 | 297

6. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: Number of participants with AESIs were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Thrombotic events and/or thrombocytopenia (defined as platelet count below the lower limit of normal [LLN] range for the testing lab) were considered to be potential AESIs.
Time Frame: Up to 6 months after the last vaccination (up to Month 18)
Population: The FAS set included all randomized participants who received at least one vaccine administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C and Mosaic gp140 | Group 2: Placebo
Number analyzed (Participants) | 1942 | 1945
Participants | 4 | 2

7. Secondary Outcome: Number of Participants With Medically-attended Adverse Events (MAAEs)
Description: Number of participants with MAAEs were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. MAAEs are defined as AEs with medically-attended visits including hospital, emergency room, urgent care clinic, or other visits to or from medical personnel for any reason.
Time Frame: From Day 1 up to Month 40
Population: The FAS set included all randomized participants who received at least one vaccine administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C and Mosaic gp140 | Group 2: Placebo
Number analyzed (Participants) | 1942 | 1945
Participants | 999 | 1002

8. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Number of participants with SAEs were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect; suspected transmission of any infectious agent via a medicinal product or medically important.
Time Frame: From Day 1 up to Month 40
Population: The FAS set included all randomized participants who received at least one vaccine administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C and Mosaic gp140 | Group 2: Placebo
Number analyzed (Participants) | 1942 | 1945
Participants | 82 | 77

9. Secondary Outcome: Number of Participants Who Discontinued the Study or Study Intervention Due to Adverse Events (AEs)
Description: Number of participants who discontinued the study or study intervention due to AEs were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Time Frame: From Day 1 up to Month 40
Population: The FAS set included all randomized participants who received at least one vaccine administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C and Mosaic gp140 | Group 2: Placebo
Number analyzed (Participants) | 1942 | 1945
Participants | 11 | 16

10. Secondary Outcome: Number of Participants With a Confirmed Human Immunodeficiency Virus (HIV)-1 Infections Diagnosed Over Time (Modified Intent-to-Treat [mITT] Set)
Description: Number of participants with a confirmed HIV-1 infections diagnosed over time (mITT set) were reported. The data represents the cumulative incidence of HIV-1 infections at specified intervals.
Time Frame: Month 0 to 24, Month 0 to 30, Month 0 to 40
Population: The mITT efficacy population included participants in the FAS who were HIV-1 uninfected at the date of the first vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C and Mosaic gp140 | Group 2: Placebo
Number analyzed (Participants) | 1940 | 1938
Participants
  Month 0 to 24 | 124 | 123
  Month 0 to 30 | 130 | 132
  Month 0 to 40 | 130 | 133

11. Secondary Outcome: Number of Participants With a Confirmed Human Immunodeficiency Virus (HIV)-1 Infections Diagnosed Over Time (Modified Intent-to-Treat-2 [mITT-2] Set)
Description: Number of participants with a confirmed HIV-1 infections diagnosed over time (mITT-2 set) were reported. The data represents the cumulative incidence of HIV-1 infections at specified intervals.
Time Frame: Month 7 to 24, Month 7 to 30, Month 7 to 40
Population: The mITT-2 efficacy population included participants in the FAS who had a negative HIV test 4 weeks post third vaccination visit (that is, at the Month 7 Visit).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C and Mosaic gp140 | Group 2: Placebo
Number analyzed (Participants) | 1812 | 1796
Participants
  Month 7 to 24 | 75 | 71
  Month 7 to 30 | 81 | 80
  Month 7 to 40 | 81 | 81

12. Secondary Outcome: Number of Participants With Confirmed Human Immunodeficiency Virus (HIV)-1 Infections Diagnosed Over Time (Modified Intent-to-Treat-3 [mITT-3] Set)
Description: Number of participants with confirmed HIV-1 infection diagnosed over time (mITT-3 set) were reported. The data represents the cumulative incidence of HIV-1 infections at specified intervals.
Time Frame: Month 7 to 24, Month 7 to 30, Month 7 to 40
Population: The mITT-3 efficacy population included participants in the FAS who had a negative HIV test 4 weeks post third vaccination visit (that is, at the Month 7 Visit) and who received all planned vaccinations at the first three vaccination visits regardless of the fact if the vaccinations were within the visit windows.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C and Mosaic gp140 | Group 2: Placebo
Number analyzed (Participants) | 1793 | 1775
Participants
  Month 7 to 24 | 75 | 71
  Month 7 to 30 | 81 | 80
  Month 7 to 40 | 81 | 81

13. Secondary Outcome: Number of Participants With Confirmed Human Immunodeficiency Virus (HIV)-1 Infections Diagnosed Over Time (Full Immunization Analysis Set [FIS])
Description: Number of participants with confirmed HIV-1 infection diagnosed over time (FIS set) were reported. The data represents the cumulative incidence of HIV-1 infections at specified intervals.
Time Frame: Month 13 to 24, Month 13 to 30, Month 13 to 40
Population: The FIS included participants in the FAS who were HIV-1 uninfected 4 weeks after the fourth vaccination visit (that is, at Month 13 Visit) and who received all planned vaccinations within the respective visit windows.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C and Mosaic gp140 | Group 2: Placebo
Number analyzed (Participants) | 1383 | 1376
Participants
  Month 13 to 24 | 22 | 22
  Month 13 to 30 | 28 | 31
  Month 13 to 40 | 28 | 32

14. Secondary Outcome: Number of Participants With Confirmed Human Immunodeficiency Virus (HIV)-1 Infections as Assessed by Demographic Characteristics: Age Groups
Description: Number of participants with confirmed HIV-1 infection as assessed by demographic characteristics: age groups was reported. Age groups included 18-20, 21-24, 25-29, 30-34, 35-44, and greater than or equal to (>=) 45 years. The data represents the cumulative incidence of HIV-1 infections at specified intervals.
Time Frame: Month 7 to 24, Month 7 to 30, Month 7 to 40
Population: The PP set included all participants in the FAS (who received at least one vaccine administration) population who had a negative HIV test 4 weeks post third vaccination visit (that is, at Month 7 Visit) and who received all planned vaccinations at the first 3 vaccination visits within the respective visit windows. Here, 'n' (number analyzed) indicated participants analyzed at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C and Mosaic gp140 | Group 2: Placebo
Number analyzed (Participants) | 1525 | 1494
Participants
  Month 7 to 24 (Age Group: 18-20 years): number analyzed (Participants) | 140 | 138
  Month 7 to 24 (Age Group: 18-20 years) | 8 | 7
  Month 7 to 24 (Age Group: 21-24 years): number analyzed (Participants) | 298 | 275
  Month 7 to 24 (Age Group: 21-24 years) | 15 | 17
  Month 7 to 24 (Age Group: 25-29 years): number analyzed (Participants) | 406 | 414
  Month 7 to 24 (Age Group: 25-29 years) | 21 | 17
  Month 7 to 24 (Age Group: 30-34 years): number analyzed (Participants) | 296 | 288
  Month 7 to 24 (Age Group: 30-34 years) | 7 | 7
  Month 7 to 24 (Age Group: 35-44 years): number analyzed (Participants) | 274 | 256
  Month 7 to 24 (Age Group: 35-44 years) | 12 | 6
  Month 7 to 24 (Age Group: >=45 years): number analyzed (Participants) | 111 | 123
  Month 7 to 24 (Age Group: >=45 years) | 2 | 4
  Month 7 to 30 (Age Group: 18-20 years): number analyzed (Participants) | 140 | 138
  Month 7 to 30 (Age Group: 18-20 years) | 9 | 10
  Month 7 to 30 (Age Group: 21-24 years): number analyzed (Participants) | 298 | 275
  Month 7 to 30 (Age Group: 21-24 years) | 18 | 17
  Month 7 to 30 (Age Group: 25-29 years): number analyzed (Participants) | 406 | 414
  Month 7 to 30 (Age Group: 25-29 years) | 22 | 21
  Month 7 to 30 (Age Group: 30-34 years): number analyzed (Participants) | 296 | 288
  Month 7 to 30 (Age Group: 30-34 years) | 8 | 8
  Month 7 to 30 (Age Group: 35-44 years): number analyzed (Participants) | 274 | 256
  Month 7 to 30 (Age Group: 35-44 years) | 12 | 7
  Month 7 to 30 (Age Group: >=45 years): number analyzed (Participants) | 111 | 123
  Month 7 to 30 (Age Group: >=45 years) | 2 | 4
  Month 7 to 40 (Age Group: 18-20 years): number analyzed (Participants) | 140 | 138
  Month 7 to 40 (Age Group: 18-20 years) | 9 | 10
  Month 7 to 40 (Age Group: 21-24 years): number analyzed (Participants) | 298 | 275
  Month 7 to 40 (Age Group: 21-24 years) | 18 | 17
  Month 7 to 40 (Age Group: 25-29 years): number analyzed (Participants) | 406 | 414
  Month 7 to 40 (Age Group: 25-29 years) | 22 | 22
  Month 7 to 40 (Age Group: 30-34 years): number analyzed (Participants) | 296 | 288
  Month 7 to 40 (Age Group: 30-34 years) | 8 | 8
  Month 7 to 40 (Age Group: 35-44 years): number analyzed (Participants) | 274 | 256
  Month 7 to 40 (Age Group: 35-44 years) | 12 | 7
  Month 7 to 40 (Age Group: >=45 years): number analyzed (Participants) | 111 | 123
  Month 7 to 40 (Age Group: >=45 years) | 2 | 4

15. Secondary Outcome: Number of Participants With Confirmed Human Immunodeficiency Virus (HIV)-1 Infections as Assessed by Demographic Characteristics: Region-Wise Enrollment
Description: Number of participants with confirmed HIV-1 infections as assessed by demographic characteristics: region-wise enrollment was reported. Regions were Latin-America (Argentina, Brazil, Mexico, and Peru), North America (Puerto Rico and United States of America), and Europe (Italy, Poland, and Spain). The data represents the cumulative incidence of HIV-1 infections at specified intervals.
Time Frame: Month 7 to 24, Month 7 to 30, Month 7 to 40
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C and Mosaic gp140 | Group 2: Placebo
Number analyzed (Participants) | 1525 | 1494
Participants
  Month 7 to 24: Latin America: number analyzed (Participants) | 1244 | 1214
  Month 7 to 24: Latin America | 63 | 54
  Month 7 to 24: North America: number analyzed (Participants) | 74 | 71
  Month 7 to 24: North America | 0 | 1
  Month 7 to 24: Europe: number analyzed (Participants) | 207 | 209
  Month 7 to 24: Europe | 2 | 3
  Month 7 to 30: Latin America: number analyzed (Participants) | 1244 | 1214
  Month 7 to 30: Latin America | 68 | 63
  Month 7 to 30: North America: number analyzed (Participants) | 74 | 71
  Month 7 to 30: North America | 0 | 1
  Month 7 to 30: Europe: number analyzed (Participants) | 207 | 209
  Month 7 to 30: Europe | 3 | 3
  Month 7 to 40: Latin America: number analyzed (Participants) | 1244 | 1214
  Month 7 to 40: Latin America | 68 | 64
  Month 7 to 40: North America: number analyzed (Participants) | 74 | 71
  Month 7 to 40: North America | 0 | 1
  Month 7 to 40: Europe: number analyzed (Participants) | 207 | 209
  Month 7 to 40: Europe | 3 | 3

16. Secondary Outcome: Number of Participants With an HIV-1 Infection by Adenovirus Serotype 26 (Ad26) at Baseline
Description: Number of participants with an HIV-1 infection by Ad26 at baseline were reported.
Time Frame: Baseline (Day 1)
Population: The immunogenicity analysis set included participants who acquired HIV-1 (case) and HIV-1 test negative (controls) that were selected for the case-control analysis. Here, 'N' (number of participants analyzed) indicates number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C and Mosaic gp140 | Group 2: Placebo
Number analyzed (Participants) | 364 | 23
Participants | 204 | 10

17. Secondary Outcome: Geometric Mean Antibody Titers For Adenovirus Serotype 26 (Ad26) as Determined by Vector Neutralization Assay (VNA)
Description: Geometric mean antibody titers for Ad26 as determined by VNA were reported.
Time Frame: From Day 1 up to Month 40
Population: The immunogenicity analysis set included participants who acquired HIV-1 (case) and HIV-1 test negative (controls) that were selected for the analysis. Here, 'N' (number of participants analyzed) indicates number of participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C and Mosaic gp140 | Group 2: Placebo
Number analyzed (Participants) | 364 | 23
Titers | 66.6 (54.1) [54.1 to 82.0] | 41.3 (16.1) [16.1 to 106.2]

18. Secondary Outcome: Number of Participants With HIV-1 Infection by Pre/Post-exposure Prophylaxis (P[r]EP) Use
Description: Number of participants with HIV-1 infection by P(r)EP use were reported. P(r)EP was assessed with a 4 item survey. Each item was measured on a scale ranging from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicating higher levels of self-efficacy. If participant showed any evidence of P(r)EP use during the period based on questionnaire responses, concomitant medications or dried blood spot analysis, the response was "yes". The data represents the cumulative incidence of HIV-1 infections at specified intervals.
Time Frame: Month 7 to 24, Month 7 to 30, Month 7 to 40
Population: The PP set included all subjects in FAS (all randomized participants who received at least one vaccine) set who had a negative HIV test 4 weeks post 3rd vaccination visit (that is, at Month 7 Visit) and who received all planned vaccinations at the first three vaccination visits within respective visit windows. Here, 'N' (number of participants analyzed) is number of participants evaluable for this outcome measure and 'n' (number analyzed) indicated participants analyzed at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C and Mosaic gp140 | Group 2: Placebo
Number analyzed (Participants) | 1525 | 1494
Participants
  Month 7 to 24: P(r)EP Use=Y: number analyzed (Participants) | 335 | 359
  Month 7 to 24: P(r)EP Use=Y | 5 | 3
  Month 7 to 24: P(r)EP Use=N: number analyzed (Participants) | 1190 | 1135
  Month 7 to 24: P(r)EP Use=N | 60 | 55
  Month 7 to 30: P(r)EP Use=Y: number analyzed (Participants) | 355 | 371
  Month 7 to 30: P(r)EP Use=Y | 5 | 5
  Month 7 to 30: P(r)EP Use=N: number analyzed (Participants) | 1170 | 1123
  Month 7 to 30: P(r)EP Use=N | 66 | 62
  Month 7 to 40: P(r)EP Use=Y: number analyzed (Participants) | 355 | 372
  Month 7 to 40: P(r)EP Use=Y | 5 | 5
  Month 7 to 40: P(r)EP Use=N: number analyzed (Participants) | 1170 | 1122
  Month 7 to 40: P(r)EP Use=N | 66 | 63

ADVERSE EVENTS:
Time Frame: Unsolicited AEs: 28 days after each vaccination (up to Day 392); Solicited AEs: 7 days after each vaccination (up to Day 371); All-cause mortality and SAE: From Day 1 up to Month 40
Description: The full analysis set (FAS) set included all randomized participants who received at least one vaccine administration.
Arm/Group | Group 1: Ad26.Mos4.HIV + Clade C and Mosaic gp140 | Group 2: Placebo
All-Cause Mortality (participants affected / at risk) | 4/1942 | 6/1945
Serious Adverse Events (participants affected / at risk) | 82/1942 | 77/1945
Other Adverse Events (participants affected / at risk) | 1687/1942 | 1348/1945
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Ad26.Mos4.HIV + Clade C and Mosaic gp140 (N=1942) | Group 2: Placebo (N=1945)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Alcoholic Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal Fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileal Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incarcerated Umbilical Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oedematous Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abdominal Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Abscess Jaw (Infections and infestations) | 1 (1) | 0 (0)
Abscess Limb (Infections and infestations) | 1 (1) | 0 (0)
Acute HIV Infection (Infections and infestations) | 1 (1) | 1 (3)
Acute Hepatitis C (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 8 (8) | 11 (11)
Bacterial Colitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 5 (5) | 2 (2)
COVID-19 Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Complicated Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Dengue Fever (Infections and infestations) | 0 (0) | 2 (2)
Fournier's Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0)
Helicobacter Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis A (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Meningitis Tuberculous (Infections and infestations) | 0 (0) | 1 (1)
Meningitis Viral (Infections and infestations) | 1 (1) | 0 (0)
Monkeypox (Infections and infestations) | 2 (2) | 1 (1)
Neurosyphilis (Infections and infestations) | 3 (3) | 0 (0)
Osteomyelitis Chronic (Infections and infestations) | 0 (0) | 1 (1)
Peritonsillar Abscess (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2)
Pulmonary Sepsis (Infections and infestations) | 3 (3) | 0 (0)
Pulmonary Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis Acute (Infections and infestations) | 0 (0) | 1 (1)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1)
Soft Tissue Infection (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous Abscess (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Hand Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint Dislocation (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Joint Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament Rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple Injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumothorax Traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post-Traumatic Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Traumatic Intracranial Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic Lung Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood Creatine Phosphokinase Increased (Investigations) | 1 (1) | 0 (0)
Diabetic Metabolic Decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Facial Asymmetry (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bone Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Head and Neck Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
T-Cell Type Acute Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Testicular Seminoma (Pure) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Nerve Compression (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Patient-Device Incompatibility (Product Issues) | 0 (0) | 1 (1)
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Behaviour Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Bipolar Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Completed Suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (2)
Depression Suicidal (Psychiatric disorders) | 0 (0) | 1 (2)
Drug Abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Drug Use Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Generalised Anxiety Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Intentional Self-Injury (Psychiatric disorders) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 1 (1) | 0 (0)
Mental Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 4 (4) | 6 (7)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus Urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal Failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary Tract Obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax Spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cellulite (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nasal Septal Operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Peripheral Venous Disease (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Ad26.Mos4.HIV + Clade C and Mosaic gp140 (N=1942) | Group 2: Placebo (N=1945)
Diarrhoea (Gastrointestinal disorders) | 51 (60) | 54 (61)
Nausea (Solicited) (Gastrointestinal disorders) | 520 (758) | 361 (552)
Vomiting (Solicited) (Gastrointestinal disorders) | 128 (154) | 85 (115)
Chills (Solicited) (General disorders) | 857 (1405) | 342 (533)
Fatigue (Solicited) (General disorders) | 1323 (3376) | 928 (2018)
Pyrexia (Solicited) (General disorders) | 400 (508) | 137 (174)
Vaccination Site Erythema (Solicited) (General disorders) | 47 (66) | 7 (7)
Vaccination Site Pain (Solicited) (General disorders) | 1519 (5543) | 695 (1521)
Vaccination Site Swelling (Solicited) (General disorders) | 89 (144) | 9 (10)
Anal Chlamydia Infection (Infections and infestations) | 22 (22) | 39 (39)
COVID-19 (Infections and infestations) | 75 (76) | 79 (81)
Gastroenteritis (Infections and infestations) | 16 (16) | 23 (23)
Influenza (Infections and infestations) | 34 (35) | 34 (38)
Nasopharyngitis (Infections and infestations) | 25 (25) | 28 (29)
Oropharyngeal Gonococcal Infection (Infections and infestations) | 27 (28) | 40 (43)
Pharyngitis (Infections and infestations) | 20 (22) | 20 (21)
Proctitis Gonococcal (Infections and infestations) | 33 (33) | 32 (33)
Syphilis (Infections and infestations) | 24 (25) | 40 (41)
Upper Respiratory Tract Infection (Infections and infestations) | 29 (31) | 27 (28)
Arthralgia (Solicited) (Musculoskeletal and connective tissue disorders) | 806 (1503) | 380 (639)
Myalgia (Solicited) (Musculoskeletal and connective tissue disorders) | 1124 (2333) | 563 (991)
Headache (Solicited) (Nervous system disorders) | 1181 (2550) | 863 (1834)
Hypertension (Vascular disorders) | 17 (18) | 24 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor and its partners for review at least 21 days before submission for publication or presentation. At the request of the sponsor and/or partners, such submission may be delayed up to 60 days. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/15/NCT03964415/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-05): https://cdn.clinicaltrials.gov/large-docs/15/NCT03964415/SAP_001.pdf